CLINICAL TRIAL: NCT06767891
Title: A Prospective, National, Multi-center, Observational Real-world Study of Acalabrutinib in Chinese MCL/CLL Patients (RESA)
Brief Title: Real-world Study of Acalabrutinib
Status: Enrolling by invitation | Type: Observational
Sponsor: Ruijin Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: ESR-22-21992
Record Dates: First submitted 2024-10-30; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-08

CONDITIONS: MCL; CLL
Keywords: Acalabrutinib; MCL; CLL

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MCL: Chinese patients with MCL treated with acalabrutinib
- CLL: Chinese patients with CLL treated with acalabrutinib

SUMMARY:
The primary purpose of this study was to describe acotinib treatment patterns among Chinese patients with CLL and MCL who received acotinib according to the label. Secondary objectives include: 1) To evaluate the safety of acotinib in Chinese patients with CLL and MCL who received acotinib according to the label. 2) Evaluate the dose of acotinib in Chinese patients with CLL and MCL who receive acotinib according to the label. 3) Describe the baseline clinical and demographic characteristics of patients with CLL and MCL who received acotinib according to the label. The exploratory objectives of the study include: 1) To describe the real-world overall survival (rwOS) of Chinese CLL and MCL patients treated with acotinib according to the label. 2) Describe the real-world clinical progression-free survival (rwPFS) of Chinese CLL and MCL patients who received acotinib according to the label. 3) Describe the real-world response rate (rwRR) in Chinese CLL and MCL patients who received acotinib according to the label.

ELIGIBILITY:
Inclusion Criteria:

* 1: Patients should be ≥18 years old at diagnosis
* 2: Diagnosed as MCL or CLL who have received at least one prior therapy and CLL patients should be enrolled after the approval of NMPA (according to Chinese label)
* 3: Eligible for acalabrutinib treatment assessed by investigators (physician's evaluation) in clinical practice
* 4: Patient/legal guardian must be able to read, understand, and sign the informed consent form (ICF)

Exclusion Criteria:

* 1: Ineligible for acalabrutinib treatment assessed by investigators (physician's evaluation)
* 2: Progression after accepting other BTKi treatment before use of acalabrutinib
* 3: Concurrent participation in another interventional clinical study
* 4: Females of childbearing potential must practice highly effective contraception during treatment of acalabrutinib, and for at least 1 week after the last dose of acalabrutinib, and have a negative urine or serum pregnancy test ≤ 7 days before the first dose of study drug(s).
* 5: No requirement to use contraception for male subjects treated with acalabrutinib. a. A sterile male is considered a highly effective contraception method for female patients. b. Males with known "low sperm counts" (consistent with "sub-fertility") are not to be considered sterile for purposes of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese MCL and CLL patients treated with acalabrutinib
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
treatment patterns | 2028/1
  Acalabrutinib treatment pattern will be summarized by the percentage of patients with acalabrutinib monotherapy and combo-therapies. Among patients with acalabrutinib combo-therapy, the frequency and percentage of patients in each categories (e.g. chemo, anti-CD20mAb, BCL2i, immunomodulator, etc.) will also be summarized. The Clopper-Pearson 95% confidence intervals (CIs) will also be presented.

SECONDARY OUTCOMES:
The percentage of patients with AEs, SAEs (safety) | 2028/1
  The percentage of patients with AEs, SAEs, will be summarized by System Organ Class and preferred term. The Clopper-Pearson 95% CIs around the incidence rate will also be reported.
posology | 2028/1
  Posology of acalabrutinib in Chinese CLL and MCL patients who received acalabrutinib according to Chinese label

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided